CLINICAL TRIAL: NCT00799058
Title: A DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED PHASE I/II TRIAL TO EVALUATE THE SAFETY OF DAPIVIRINE GEL 4759, 0.05% 2.5g AND DAPIVIRINE GEL 4789, 0.05% 2.5g FORMULATIONS AS COMPARED TO THE VAGINAL HEC-BASED UNIVERSAL PLACEBO GEL, 2.5g IN HEALTHY HIV-NEGATIVE WOMEN
Brief Title: A Safety Study of Two Dapivirine (TMC120) Vaginal Gels in the United States
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 020
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: HIV-1 Infections
Keywords: HIV-1 infections
MeSH Terms: interventions — Dapivirine

STUDY DESIGN:
Intervention Model Description: All enrolled participants will apply gel on a daily basis for 12 weeks, with clinical follow-up visits at weeks 2,4,8 and 12 to monitor safety and acceptability, and a final visit 4 weeks post gel discontinuation (Visit 6, week 16) Dapivirine concentration will be measured in blood and vaginal fluid and cervical tissue.
Who Masked: Participant, Investigator
Masking Description: Potential participants who provide inform consent will be invited to screen for the trial. All participants who consent to participate in the trial and meet specified inclusion/exclusion criteria will be invited to enrol. At enrolment women will be randomly assigned in a 1:1:1 ratio to one of three groups.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dapivirine gel 4789 (Active Comparator): will be applied by participants once daily for 12-weeks treatment period
  Interventions: Drug: dapivirine 4789
- dapivirine gel 4759 (Active Comparator): Will be applied by participants once daily for12-weeks treatment period
  Interventions: Drug: dapivirine gel 4759
- HEC-based placebo gel, 2.5g containing no Dapivirine (Placebo Comparator): Will be applied once daily for 12-weeks treatment period
  Interventions: Drug: Drug placebo

INTERVENTIONS:
Drug: dapivirine 4789 — dapivirine gel 4789, 0.05%, 2.5g applied once daily
  Other Names: TMC120
  Arms: dapivirine gel 4789
Drug: dapivirine gel 4759 — dapivirine gel 4759, 0.05%, 2.5g applied once daily
  Other Names: TMC120
  Arms: dapivirine gel 4759
Drug: Drug placebo — HEC-based universal placebo gel, 2.5g applied once daily
  Other Names: HEC-based placebo gel, 2.5g
  Arms: HEC-based placebo gel, 2.5g containing no Dapivirine

SUMMARY:
A double-blind, randomized, placebo-controlled Phase I/II trial to evaluate the safety of dapivirine Gel 4759, 0.05% 2.5 g and dapivirine Gel 4789, 0.05% 2.5 g formulations as compared to the vaginal HEC-based Universal placebo gel, 2.5 g in healthy HIV-negative women

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled trial, to be conducted over 10 months at five research centers in the USA among 180 healthy, sexually active women, to assess the safety and acceptability of dapivirine Gel 4759, 0.05% 2.5 g, and dapivirine Gel 4789, 0.05% 2.5 g, both vaginal microbicides containing dapivirine, compared to the vaginal HEC-based Universal placebo gel, 2.5 g, containing no active ingredient, used once daily for a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 to 40 years of age inclusive who can give written informed consent
2. Available for all visits and consent to follow all procedures scheduled for the trial
3. Healthy and self-reported sexually active
4. HIV-negative as determined by an HIV test at time of enrollment
5. Willing to be on a stable form of contraception
6. In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle
7. Upon pelvic/speculum examination and colposcopy at the enrollment visit, the cervix and vagina appear normal as determined by qualified research center staff
8. Asymptomatic for genital infections at the time of enrollment
9. Willing to refrain from use of vaginal products or objects for 14 days prior to enrollment and for the duration of the trial.
10. Documentation of no abnormality on Pap smear within 90 days prior to randomization;
11. Willing to answer acceptability and adherence questionnaires throughout the trial
12. Willing to refrain from participation in any other research trial for the duration of this trial
13. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures
14. Willing to abstain from all the following criteria beginning 48 hours prior to each trial visit:

    * Vaginal intercourse
    * Oral contact with her genitalia
    * Internal vaginal washing
    * Penetration of the vagina by fingers, sex toys, or any other objects, including medications
15. Willing to abstain from all of the following for 3 days after biopsy procedures:

    * Vaginal intercourse
    * Oral contact with her genitalia
    * Internal vaginal washing
    * Penetration of the vagina by fingers, sex toys, or any other objects, including medications

Exclusion Criteria:

1. Currently pregnant or having had their last pregnancy outcome within 3 months prior to screening
2. Currently breast-feeding, or having breastfed within 3 months prior to screening
3. Receipt of any investigational agent within 60 days prior to screening
4. Previously participated in any HIV vaccine trial
5. Untreated urogenital infections within 2 weeks prior to enrollment
6. Presence of any abnormal physical finding on the vulva, vaginal walls or cervix during pelvic/speculum examination and/or colposcopy
7. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, or urethral obstruction
8. Pap smear result at screening that requires cryotherapy, biopsy or treatment (other than for infection)
9. History of symptomatic or asymptomatic HSV-2
10. Any Grade 2, 3 or 4 hematology, chemistry or urinalysis laboratory abnormality at baseline
11. Unexplained, undiagnosed abnormal bleeding per vagina during or following vaginal intercourse; or urogenital surgery within 90 days prior to enrollment
12. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex
13. Any serious acute, chronic or progressive disease
14. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2009-07-06 (Actual); Primary Completion 2011-01-08 (Actual); Study Completion 2011-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Annalene Nel, Study Chair — International Partnership for Microbicides
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Alabama Microbicide Clinical Research Site (AMCRS), Birmingham, Alabama
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Illinois at Chicago, Chicago, Illinois
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland
  - Albert Einstein College of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 180 women (35-50 per RC) were scheduled to be enrolled at 5 research centers in the USA. However, following IPM's decision to give priority to development of the dapivirine vaginal ring above that of dapivirine vaginal gel, the Sponsor decided to stop enrollment into IPM 020 trial after 128 participants were randomized. It was determined that the number of participants already enrolled were sufficient to allow for meaningful analysis of the data. Total trial duration was 18 months.
Period: Overall Study
Arm/Group | Dapivirine Gel 4789 | Dapivirine Gel 4759 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
Started | 43 | 43 | 42
Completed | 33 | 34 | 36
Not Completed | 10 | 9 | 6
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Not adherent | 3 | 2 | 1
Not completed — discontinued use of IP due to AE, but completed visits | 0 | 0 | 1
Not completed — IP dispensing error | 1 | 0 | 0
Not completed — not enough IP to complete trial due to IP dispending error | 0 | 1 | 0
Not completed — IP discontinued too long during BV treatment | 1 | 0 | 0
Not completed — lost 2 IP kits and did not have enough remaining to complete trial | 0 | 0 | 1
Not completed — participant did not attend clinic visit 6 (final visit) | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy, sexually active, HIV-negative women
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine | Total
Number analyzed (Participants) | 43 | 43 | 42 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.9) | 27.5 (5.5) | 27.5 (5.5) | 27.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 42 | 128
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 10 | 9 | 4 | 23
  Black or African American | 16 | 16 | 15 | 47
  White | 17 | 14 | 18 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 42 | 128
Married [Count of Participants; unit: Participants] | 9 | 7 | 12 | 28
In a relationship with one partner, not married [Count of Participants; unit: Participants] | 35 | 38 | 29 | 102
Cohabitating with main partner [Count of Participants; unit: Participants] | 9 | 16 | 12 | 37
In a relationship with multiple partners [Count of Participants; unit: Participants] | 1 | 1 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] | 163.7 (6.8) | 163.5 (7.4) | 161.4 (8.9) | 162.9 (7.8)
Weight [Mean (Standard Deviation); unit: kg] | 77.0 (17.5) | 73.3 (14.9) | 69.2 (18.8) | 73.2 (17.3)
BMI [Mean (Standard Deviation); unit: kg/(m^2)] | 28.7 (6.3) | 27.5 (5.9) | 26.5 (6.1) | 27.6 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Women With the Composite Endpoint of Abnormal Safety Findings.
Description: A composite endpoint was defined as the percentage of participants with any post-baseline abnormal finding from pelvic/speculum examination, colposcopy finding, STI diagnoses, laboratory test of DAIDS grade 3 or higher and any product-related AE.
  DAIDS severity grades are defined as follows:
  Grade 1 = mild Grade 2 = moderate Grade 3 = severe Grade 4 = potentially life-threatening Grade 5 = death
Time Frame: 12 weeks
Population: The ITT population included all trial participants who were randomized to one of the three treatment groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
Number analyzed (Participants) | 43 | 43 | 42
Participants | 23 | 28 | 28

2. Secondary Outcome: Changes in the Vaginal Flora
Description: Cervicovaginal fluid specimens will be obtained to determine vaginal flora before first gel application and at Visits 3, 5, and 6. Appropriate statistical analyses incorporating repeated measures will be used to assess the changes in the vaginal flora in women using Dapivirine Gel 4759, 0.05% 2.5g, Dapivirine Gel 4789, 0.05% 2.5g or the vaginal HEC-based universal placebo gel, 2.5g.
  Nugent scores were used to assess changes in vaginal flora, and were categorized into three levels: (1) negative for BV (score: 0-3); (2) altered vaginal flora (score: 4-6); and (3) BV (score: 7-10).
Time Frame: 16 weeks
Population: All participants who were assigned to a treatment group were analyzed as members of the group to which they were randomized, regardless of adherence to the planned course of treatment.
  Results are reported for participants who provided vaginal samples.
Measure: Number; unit: percentage of participants with data
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
Number analyzed (Participants) | 43 | 43 | 42
percentage of participants with data
  Week 0 : Normal Flora (0-3): number analyzed (Participants) | 28 | 26 | 23
  Week 0 : Normal Flora (0-3) | 66.7 | 60.5 | 54.8
  Week 0 : Altered Flora (4-6): number analyzed (Participants) | 6 | 5 | 10
  Week 0 : Altered Flora (4-6) | 14.3 | 11.6 | 23.8
  Week 0 : Abnormal Flora (7 or more): number analyzed (Participants) | 8 | 12 | 9
  Week 0 : Abnormal Flora (7 or more) | 19.0 | 27.9 | 21.4
  Week 4 : Normal Flora (0-3): number analyzed (Participants) | 25 | 22 | 27
  Week 4 : Normal Flora (0-3) | 67.6 | 55.0 | 65.9
  Week 4 : Altered Flora (4-6): number analyzed (Participants) | 3 | 5 | 8
  Week 4 : Altered Flora (4-6) | 8.1 | 12.5 | 19.5
  Week 4 : Abnormal Flora (7 or more): number analyzed (Participants) | 9 | 13 | 6
  Week 4 : Abnormal Flora (7 or more) | 24.3 | 32.5 | 14.6
  Week 12: Normal Flora (0-3): number analyzed (Participants) | 21 | 23 | 22
  Week 12: Normal Flora (0-3) | 61.8 | 65.7 | 59.5
  Week 12: Altered Flora (4-6): number analyzed (Participants) | 8 | 7 | 9
  Week 12: Altered Flora (4-6) | 23.5 | 20.0 | 24.3
  Week 12: Abnormal Flora (7 or more): number analyzed (Participants) | 5 | 5 | 6
  Week 12: Abnormal Flora (7 or more) | 14.7 | 14.3 | 16.2
  Week 16 (Follow-up after IP discontinuation): Normal Flora (0-3): number analyzed (Participants) | 24 | 22 | 24
  Week 16 (Follow-up after IP discontinuation): Normal Flora (0-3) | 70.6 | 66.7 | 64.9
  Week 16 (Follow-up after IP discontinuation): Altered Flora (4-6): number analyzed (Participants) | 1 | 6 | 7
  Week 16 (Follow-up after IP discontinuation): Altered Flora (4-6) | 2.9 | 18.2 | 18.9
  Week 16 (Follow-up after IP discontinuation): Abnormal Flora (7 or more): number analyzed (Participants) | 9 | 5 | 6
  Week 16 (Follow-up after IP discontinuation): Abnormal Flora (7 or more) | 26.5 | 15.2 | 16.2

3. Secondary Outcome: The Distribution of Dapivirine Levels Observed in Plasma Samples at Each Specified Time Point
Description: Dapivirine levels observed in plasma will be summarized using simple descriptive statistics.
Time Frame: 12 weeks
Population: The PK analysis population included all participants who received at least one dose of the active IP and for whom at least one plasma, vaginal fluid or cervical tissue sample was taken.
  Results are provided for participants for whom samples were available.
Measure: Mean (Standard Deviation); unit: picograms/mililiter
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789
Number analyzed (Participants) | 43 | 43
picograms/mililiter
  Week 2: number analyzed (Participants) | 37 | 36
  Week 2 | 536.8 (297.2) | 475.8 (272.2)
  Week 4: number analyzed (Participants) | 33 | 37
  Week 4 | 599.5 (423.1) | 446.1 (272.2)
  Week 8: number analyzed (Participants) | 28 | 31
  Week 8 | 572.6 (377.5) | 432.6 (276.8)
  Week 12: number analyzed (Participants) | 30 | 33
  Week 12 | 519.1 (351.3) | 366.1 (329.6)

4. Secondary Outcome: The Adherence to Once Daily Application of a Vaginal Microbicide Gel Over a 12-week Period in Healthy, Sexually Active, HIV-negative Women
Description: Adherence is defined as the percentage of participants who used the gel each day of the preceding 14 days, based on participant self reports.
Time Frame: 12 weeks
Population: The ITT population included all trial participants who were randomized to one of the three treatment groups.
  Results are provided for participants who reported adherence information.
Measure: Number; unit: percentage of participants with data
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
Number analyzed (Participants) | 39 | 41 | 41
percentage of participants with data | 74 | 73 | 71

5. Secondary Outcome: Changes in the Vaginal pH
Description: Cervicovaginal fluid specimens will be obtained to determine vaginal pH before first gel application and at screening, enrolment and visit 5 (week 12). Appropriate statistical analyses incorporating repeated measures will be used to assess the changes in the vaginal pH in women using Dapivirine Gel 4759, 0.05% 2.5g, Dapivirine Gel 4789, 0.05% 2.5g or the vaginal HEC-based universal placebo gel, 2.5g.
Time Frame: 12 weeks
Population: All participants who were assigned to a treatment group were analyzed as members of the group to which they were randomized, regardless of adherence to the planned course of treatment.
Measure: Mean (Standard Deviation); unit: Vaginal pH
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
Number analyzed (Participants) | 43 | 43 | 42
Vaginal pH
  Screening (Week 0) | 4.46 (0.53) | 4.55 (0.63) | 4.55 (0.95)
  Visit 1 (Enrollment) | 4.45 (0.52) | 4.48 (0.5) | 4.3 (0.43)
  Visit 5 (Week 12) | 4.4 (0.46) | 4.44 (0.61) | 4.38 (0.47)

6. Secondary Outcome: The Distribution of Dapivirine Levels Observed in Vaginal Fluid at Each Specified Time Point.
Description: The distribution of dapivirine levels observed in each type of sample will be summarized using simple descriptive statistics. In addition, the proportion of women with detectable dapivirine concentrations will be calculated for each type of sample at each collection time point. Exploratory analyses of dapivirine concentration data will also be performed to take into account information reported in a diary regarding menses and tampon use throughout the trial.
Time Frame: 12 weeks. Measured at 2, 4, and 8 weeks post-enrolment and at one of these at week 12; 24, 48, or 72 hours after gel discontinuation. (Participants were randomized to have vaginal fluid samples collected at one of these visits (5a, 5b, or 5c).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789
Number analyzed (Participants) | 43 | 43
nanogram/milliliter
  Visit 2 (2 weeks post-enrollment): number analyzed (Participants) | 36 | 35
  Visit 2 (2 weeks post-enrollment) | 467.1 (579.8) | 880.7 (1924)
  Visit 3 (4 weeks post-enrolment): number analyzed (Participants) | 33 | 37
  Visit 3 (4 weeks post-enrolment) | 347.8 (351.9) | 462.6 (590.0)
  Visit 4 (8 weeks post-enrolment): number analyzed (Participants) | 28 | 31
  Visit 4 (8 weeks post-enrolment) | 526.9 (580.1) | 298.1 (151)
  Visit 5a (24 hours after gel discontinuation): number analyzed (Participants) | 10 | 17
  Visit 5a (24 hours after gel discontinuation) | 192.0 (186.7) | 680.0 (1775)
  Visit 5b (48 hours after gel discontinuation): number analyzed (Participants) | 9 | 9
  Visit 5b (48 hours after gel discontinuation) | 98.63 (180.3) | 164.0 (233.1)
  Visit 5c (72 hours after gel discontinuation): number analyzed (Participants) | 9 | 7
  Visit 5c (72 hours after gel discontinuation) | 177.0 (304.9) | 245.6 (230.7)

7. Secondary Outcome: The Distribution of Dapivirine Levels Observed in Vaginal Tissue at Each Specified Time Point.
Description: The distribution of dapivirine levels observed in vaginal tissue sample will be summarized using simple descriptive statistics.
Time Frame: as for outcome 6
Population: The PK analysis population included all participants who received at least one dose of the active IP and for whom at least one plasma, vaginal fluid or cervical tissue sample was taken.
Measure: Mean (Standard Deviation); unit: nanogram/gram
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789
Number analyzed (Participants) | 28 | 32
nanogram/gram
  Visit 5a (24 hours after gel discontinuation): number analyzed (Participants) | 10 | 17
  Visit 5a (24 hours after gel discontinuation) | 3518 (3579) | 9343 (18980)
  Visit 5b (48 hours after gel discontinuation): number analyzed (Participants) | 9 | 8
  Visit 5b (48 hours after gel discontinuation) | 841.0 (1582) | 1150 (1184)
  Visit 5c (72 hours after gel discontinuation): number analyzed (Participants) | 9 | 7
  Visit 5c (72 hours after gel discontinuation) | 4781 (9161) | 1142 (1337)

8. Secondary Outcome: Acceptability of Once Daily Application of a Vaginal Microbicide Gel Over a 12-week Period in Healthy, Sexually Active, HIV-negative Women
Description: Acceptability was assessed as the percentage of participants at week 12 who were willing to use the gel every day if proven to prevent HIV.
Time Frame: 12 weeks
Population: The ITT population included all trial participants who were randomized to one of the three treatment groups.
  Results are reported for participants who provided questionnaire responses.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Gel 4789 | Dapivirine Gel 4759 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
Number analyzed (Participants) | 40 | 41 | 40
Participants | 24 | 25 | 29

ADVERSE EVENTS:
Time Frame: Trial duration: 18 months The maximum period of gel exposure in all three treatment groups was 12 weeks.
Arm/Group | Dapivirine Gel 4759 | Dapivirine Gel 4789 | HEC-based Placebo Gel, 2.5g Containing no Dapivirine
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/43 | 2/42
Other Adverse Events (participants affected / at risk) | 30/43 | 34/43 | 35/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Gel 4759 (N=43) | Dapivirine Gel 4789 (N=43) | HEC-based Placebo Gel, 2.5g Containing no Dapivirine (N=42)
Cellulitis of the left breast (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Gel 4759 (N=43) | Dapivirine Gel 4789 (N=43) | HEC-based Placebo Gel, 2.5g Containing no Dapivirine (N=42)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal Pain Lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Gonorrhoea (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Vaginal candidiasis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 7 (7) | 15 (15) | 5 (5)
Vulvovaginal myotic infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)
Cervix erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 3 (3)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Concluding a general trend in vaginal fluid data is, however, difficult as overall individual fluid levels for the two gel formulations were in the same range and differences based on median values were not consistent across visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No